CLINICAL TRIAL: NCT04597788
Title: The Role of Protein Supplemented Very Low Calorie Medical Meals on Weight and Metabolic Changes Among People With Obesity: a Randomized Controlled Trial
Brief Title: Efficacy of Protein Supplemented Very Low Calorie Meals on Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2004-604-003
Record Dates: First submitted 2020-09-03; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Sarcopenic Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein supplemented very low calorie diet program (Experimental): The lifestyle intervention using protein supplemented very low calorie meals will be implemented with individual counseling sessions for 12 months. Initial intensive weight loss stage will be delivered during the first 4 month period with total meal replacement to partial meal replacement using protein supplemented very low calorie meals. During the weight loss maintenance stage, regular intermittent very low calorie meal replacement one week per month will be delivered for the entire period. Mobile counseling will be offered to help patients achieve weight loss as well as weight loss maintenance.
  Interventions: Other: Protein supplemented very low calorie diet program
- Conventional low calorie diet program (Active Comparator): The conventional low calorie diet program will be offered to participants assigned to control group using educational material and individual counseling sessions for 12 months. Mobile counseling will be also offered for weight loss and weight loss maintenance.
  Interventions: Other: Conventional low calorie diet program

INTERVENTIONS:
Other: Protein supplemented very low calorie diet program — Protein supplemented very low calorie meal is a shake-type meal replacement with total calories of 600 to 800 calories per day and proteins provided at 1.2g of ideal body weight per day. The four-month, very low calorie diet program schedule will be as follows. In the first two weeks, all three meals are replaced, followed by two meals replaced and one meal in food in the next six weeks, and one meal replacement is recommended for the next eight weeks. For the next eight months, the intermittent very low calorie meal replacements will be provided regularly for one week a month. If a subject gains weight more than 2kg, he or she will have an additional 1 week of two meal replacements, and if a subject gains weight more than 4kg, he or she should have an additional 2 weeks of replacement.
  Individual sessions will be held 11 times during the study. Mobile counseling with dietitians or nurses will be offered to help subjects lose weight and maintain weight loss.
  Arms: Protein supplemented very low calorie diet program
Other: Conventional low calorie diet program — Low calorie diet consists of 1200 to 1500 calories will be educated and lifestyle modification will be encouraged for participants in control group. Educational materials as well as recipes for low calorie diet will be provided in individual sessions. Mobile counseling will also be offered for sticking to the diet program.
  Arms: Conventional low calorie diet program

SUMMARY:
This randomized clinical trial will evaluate the efficacy and safety of protein supplemented very low calorie meals on weight loss and weight loss maintenance among people with obesity.

DETAILED DESCRIPTION:
Approximately 30% of the Korean population has obesity or abdominal obesity and is often accompanied by obesity related complications such as cardiovascular disease, diabetes, osteoarthritis and even some types of cancer. However, there are not many lifestyle modification treatments available that have long-term effects other than drugs and surgical treatments in the management of obesity.

Preserving muscle mass should also be considered in weight loss especially for elderly adults with obesity, because decreased muscle mass and strength can negatively affect morbidity and mortality in the elderly.

Therefore, the investigators want to evaluate the effectiveness and safety of the protein supplemented very low calorie meals on weight loss, body composition as well as metabolic changes compared with traditional low calorie low fat diet in people with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI ) more than 25 kg/m2 or
* Waist circumference more than 90 cm in men or 85 cm in women

Exclusion Criteria:

* History of treatment with anti-obesity drugs or participation in another weight loss program in previous 6 months
* Weight changes more than 3 kg during the 6 months before participation
* Unstable cardiovascular events during the 6 months before participation
* Uncontrolled mood disorder
* History of eating disorder
* History of alcohol use disorder
* History of gallstone
* Chronic renal failure (estimated glomerular filtration less than 30 ml/min)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-11-16 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in weight | 12 months
  Changes of weight loss from the baseline expressed as kg

SECONDARY OUTCOMES:
Changes in body composition | 12 months
  Changes in muscle mass and fat mass from the baseline expressed as kg using bioelectrial impedance analysis (Inbody Co., Seoul, Korea)
Changes in systolic and diastolic blood pressure | 12 months
  Changes in systolic and diastolic blood pressure from the baseline expressed as mmHg
Changes in triglyceride | 12 months
  Changes in triglyceride from the baseline expressed as mg/dL
Changes in glucose | 12 months
  Changes in glucose from the baseline expressed as mg/dL
Changes in high density lipoprotein (HDL) Cholesterol | 12 months
  Changes in HDL cholesterol from the baseline expressed as mg/dL
Changes in low density lipoprotein (LDL) Cholesterol | 12 months
  Changes in LDL cholesterol from the baseline expressed as mg/dL
Changes in liver enzyme | 12 months
  Changes in aspartate and alanine aminotransferase, gamma glutamyltransferase (AST and ALT, GGT) from the baseline expressed as IU/L
Changes in insulin resistance | 12 months
  Changes in insulin resistance using the homeostatic model assessment for insulin resistance (HOMA-IR) as HOMA-IR =insulin(uIU/ml) * fasting glucose (mg/dL)*0.05551/22.5
Changes in obesity related quality of life | 12 months
  Changes in Korean version of obesity related quality of life scales (published in Korean Society for the Study of Obesity 2003;12(4):280-293 )

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Cho E, Kim S, Kim HJ, Cho B, Park JH, Kwon H, Kim JY, Go Y, Kang DG, Shin E, Lee S, Gil S, Kim H, Ahn J, Kim JY, Jung W, Go E. Effectiveness of a protein-supplemented very-low-calorie diet program for weight loss: a randomized controlled trial in South Korea. Front Nutr. 2024 Sep 12;11:1370737. doi: 10.3389/fnut.2024.1370737. eCollection 2024. PMID 39328464